CLINICAL TRIAL: NCT03265353
Title: Vascular Effects of Dietary Potassium in Humans
Brief Title: Vascular Effects of Dietary Potassium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 487998-8
Record Dates: First submitted 2017-08-25; First posted 2017-08-29 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Cardiovascular Risk Factor
Keywords: Potassium; Sodium; Vascular function

STUDY DESIGN:
Intervention Model Description: All participants will complete each arm. It is a crossover, randomized design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Moderate Potassium/Low Sodium Diet (Other): Vascular function will be assessed at both the conduit artery and microvascular level after 7 days of the moderate potassium/low sodium diet.
  Interventions: Other: Moderate Potassium/Low Sodium Diet
- Moderate Potassium/High Sodium Diet (Other): Vascular function will be assessed at both the conduit artery and microvascular level after 7 days of the moderate potassium/high sodium diet.
  Interventions: Other: Moderate Potassium/High Sodium Diet
- High Potassium/High Sodium Diet (Other): Vascular function will be assessed at both the conduit artery and microvascular level after 7 days of the high potassium/high sodium diet.
  Interventions: Other: High Potassium/High Sodium Diet

INTERVENTIONS:
Other: Moderate Potassium/Low Sodium Diet — 7 days of the prescribed diet
  Arms: Moderate Potassium/Low Sodium Diet
Other: Moderate Potassium/High Sodium Diet — 7 days of the prescribed diet
  Arms: Moderate Potassium/High Sodium Diet
Other: High Potassium/High Sodium Diet — 7 days of the prescribed diet
  Arms: High Potassium/High Sodium Diet

SUMMARY:
The purpose of this study is to determine if dietary potassium can attenuate the deleterious effects of high sodium on blood vessel function in healthy, salt-resistant participants.

DETAILED DESCRIPTION:
Cardiovascular disease remains a major Public Health problem in the U.S. and is the result of diseases such as atherosclerosis and high blood pressure (BP). Several dietary factors have been implicated as risk factors including high sodium and low potassium diets. Indeed, it is well known that excess sodium can increase BP while potassium rich diets have BP lowering properties. While the role of these two nutrients on BP is widely accepted, their impact on the vasculature has received less attention. Endothelial dysfunction, characterized by impaired dilation is an important non-traditional risk factor for atherosclerosis. Data in animal models suggest that salt loading, independent of changes in BP, results in endothelial dysfunction while evidence is mounting that potassium may be beneficial to vascular health. Further, potassium may be more effective in the presence of high sodium however the role of potassium in protecting the vasculature from a high sodium diet in salt-resistant adults has not been explored. A potential mechanism responsible for sodium induced vascular dysfunction is overproduction of reactive oxygen species resulting in reduced nitric oxide (NO) production/ bioavailability. It has been suggested that potassium can counteract sodium's effect by reducing ROS. The central hypothesis is that potassium can protect against the deleterious effects of high sodium on the vasculature by reducing oxidative stress and preserving NO. In this grant, the investigators propose to use a 21-day controlled feeding study to compare the effects of a high sodium diet (300 mmol) combined with either a high (120 mmol) or moderate (65 mmol) amount of potassium and low sodium (50 mmol) combined with moderate potassium (crossover design, diet order sequence randomized) on 2 levels of the vasculature, conduit artery and microvasculature. These experiments will be performed in salt-resistant participants to study the vascular effects alone, independent of changes in BP.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* normal blood pressure

Exclusion Criteria:

* hypertension
* history of heart disease
* diabetes
* kidney disease
* obese (BMI ≥30)
* significant weight changes in the last 6 months
* use of tobacco products
* pregnant
* on a special diet (gluten free; vegan)
* take any medications for the above conditions
* endurance trained athletes

Ages: 22 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2013-07-25 (Actual); Primary Completion 2019-09-22 (Actual); Study Completion 2019-09-22 (Actual)

PRIMARY OUTCOMES:
Conduit artery endothelial-dependent dilation | on the 7th day of each diet
  The change in flow-mediated dilation (FMD) between the 3 diets as assessed by brachial artery FMD

OTHER OUTCOMES:
Arterial Stiffness | on 7th day of each diet
  Assessed by carotid to femoral artery pulse wave velocity
Wave reflection | on 7th day of each diet
  Assessed by augmentation index
Endothelial cell expression of oxidative stress marker | on the 7th day of each diet
  Assessed in venous endothelial cells from participants.
Ambulatory blood pressure | 7 days
  Assessed by 24 hr ambulatory blood pressure monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon L Lennon, PhD, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: Undecided